CLINICAL TRIAL: NCT01573780
Title: A Phase I Study of TL32711 In Combination With Gemcitabine in Patients With Advanced Solid Tumors
Brief Title: Gemcitabine Hydrochloride and Smac Mimetic TL32711 in Treating Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor did not have funds to continue study
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 210811; NCI-2012-00202 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-13; First posted 2012-04-10 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — birinapant; Gemcitabine; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes and smac mimetic TL32711 IV over 30 minutes once weekly for 2 weeks. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Smac mimetic TL32711; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: biopsy

INTERVENTIONS:
Drug: Smac mimetic TL32711 — Given IV
  Other Names: TL32711
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies

SUMMARY:
The purpose of this study is to determine the dose of smac mimetic TL32711 that is safe and tolerated when given with gemcitabine hydrochloride to patients with advanced cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and recommended Phase II dose of TL32711 (smac mimetic TL32711) in combination with gemcitabine (gemcitabine hydrochloride) in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To determine the toxicity and safety profile of TL32711 in combination with gemcitabine in patients with advanced solid tumors.

II. To determine the pharmacokinetic profile of TL32711 and gemcitabine when administered in combination.

III. To determine the preliminary efficacy of the study combination in patients with advanced solid tumors.

IV. To determine the relationship between predictive biomarkers and clinical activity using archival tumor tissue samples for biomarker analysis.

OUTLINE: This is a dose-escalation study of smac mimetic TL32711.

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes and smac mimetic TL32711 IV over 30 minutes once weekly for 2 weeks. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumors that are advanced or metastatic that gemcitabine-based treatment is considered standard therapy
* Patient must consent to the use of their archival tumor tissue for protocol use if available
* Patient with at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 that has not been previously irradiated
* Eastern Cooperative Oncology Group (ECOG) Performance Status =< 1
* Life expectancy >= 3 months
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (system international [SI] units 1.5 x 10^6/L)
* Platelets >= 100,000 cells/m^3 (SI units 100 x 10^6/L)
* Hemoglobin >= 9.0 g/dL (SI units 90 g/L) (in the absence of transfusion within 24 hours prior to dosing)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGPT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3 x Upper Limit of Normal (ULN); In patients with known hepatic involvement, AST and ALT < 5 x ULN are allowed
* Total bilirubin =< 1.5 x ULN; in patients with known hepatic involvement, total bilirubin =< 1.5 x ULN is allowed
* Serum creatinine =< 1.5 x ULN, or 24-hr urine creatinine clearance calculation >= 60 mL/min
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Ability to understand and willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study specific procedures
* Women of childbearing potential must have a negative serum pregnancy test at screening and negative (serum or urine) pregnancy test within 48 hours prior to the first dose of the first cycle of study treatment
* Women of childbearing potential must agree to use 2 methods of adequate contraception (i.e., hormonal and barrier method) prior to enrollment, during the study, and for a period of 30 days following the last dose of study drug(s); males who are sexually active must agree to use a condom during the study for a period of 30 days following the last dose of study drug(s), and if their partner is of childbearing potential, she must agree to use a secondary method of contraception (i.e., hormonal, intrauterine device, barrier) during the study and for a period of 30 days following the last dose of study drug(s)

Exclusion Criteria:

* Patients who have receive recent anti-cancer therapy defined by:
* Chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosourea, mitomycin-C, targeted therapy and radiation) =< 4 weeks prior to starting study drug, or who have not recovered from side effects of such therapy
* Last administration of nitrosourea or mitomycin-C =< 6 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy; or
* Targeted therapy (e.g. sunitinib, sorafenib, pazopanib) =< 2 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy; or
* Radiotherapy =< 4 weeks prior to starting study drug, or =< 2 weeks prior to starting study drug in the case of localized radiotherapy (e.g. for analgesic purpose or for lytic lesions at risk of fracture), or who have not recovered from radiotherapy toxicities
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury =< 4 weeks prior to starting study treatment, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device =< 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Uncontrolled concurrent illness, including but not limited to ongoing or active serious infection requiring systemic antimicrobials (within 2 weeks prior to first dose of TL32711), arterial hypertension (> 160/100 mm/Hg on antihypertensive medications), uncontrolled endocrine diseases, altered mental status or psychiatric illness/social situations that would limit compliance with protocol requirements and/or obscure study results
* Known or suspected diagnosis of human immunodeficiency virus (HIV) or chronic active Hepatitis B or C; viral testing is not required
* Inability to start prophylactic anti-viral medication
* Clinically significant pulmonary illness resulting in Grade >= 2 hypoxia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE, v4]) or any requirement for supplemental oxygen, or pulse oximetry less than 90% saturation on room air
* Symptomatic or uncontrolled brain metastases requiring current treatment (less than 4 weeks from last cranial radiation or 4 weeks from last steroids)
* Impaired cardiac function or clinically significant cardiac disease including the following:

  * Clinically significant arrhythmias (except chronic well controlled atrial fibrillation)
  * New York Heart Association (NYHA) grade II, III, or IV congestive heart failure
  * Angina pectoris =< 6 months prior to dosing with TL32711
  * Myocardial infarction within the last 12 months prior to dosing with TL32711
* QT interval corrected for heart rate (QTc) > 480 msec (including patients on medication); patients with a ventricular pacemaker for whom QT interval is not measurable may be eligible for enrollment after consultation with the Sponsor and the documentation of approval
* Ongoing auto-immune disease or with history of an auto-immune disease within the past 5 years; a patient with a history of auto-immune disease that is currently in remission must not be receiving medication designed to control the disease and must not have experienced an exacerbation of the disease requiring treatment with immunomodulatory agents in the last 5 years; auto-immune disease includes but are not limited to systemic lupus erythematosis, scleroderma, rheumatoid arthritis, psoriasis, psoriatic arthritis, ulcerative colitis and regional enteritis (Crohn's disease)
* Systemic or chronic topical corticosteroids or immunosuppressive therapy within 4 weeks prior to study entry or anticipated need of systemic corticosteroids or immunosuppressive therapy during study participation
* Patients with a healing or open wound
* Skin lesions of Grade >= 2 severity (NCI CTCAE v4), except alopecia
* Lack of recovery or prior adverse events to Grade =< 1 severity (NCI CTCAE v4) (except alopecia) due to medications administered prior to the first dose of TL32711
* Patients with prior history of Bell's Palsy
* Any other condition or finding that in the opinion of the investigator may render the patient at excessive risk for treatment complications or may not be able to provide evaluable outcome information
* Pregnant or breast-feeding women
* Known allergy to any of the formulation components of TL32711 including citric acid monohydrate, sodium citrate dehydrate, and sodium chloride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
MTD of smac mimetic TL32711 | During the first course (21 days)
  Defined as the highest dose level at which less than 2 of 6 patients experience study treatment-related dose-limiting toxicity. Summarized with frequencies and descriptive measures, and tabulated according to body system, severity and relation to treatment.

SECONDARY OUTCOMES:
Overall toxicity profile characterized by type, frequency, severity (according to the NCI CTCAE version 4.0), timing, seriousness, and relationship to study treatment | Up to 4 weeks post-treatment
  Summarized with frequencies and descriptive measures, and tabulated according to body system, severity and relation to treatment.
Response rates according to the RECIST v1.1 (solid tumor/dose-finding cohort) | Up to 4 weeks post-treatment
  Data presented in tabular format and summarized descriptively.
Progression-free survival | Up to 2 years
Plasma pharmacokinetic parameters of smac mimetic TL32711, gemcitabine hydrochloride and its metabolites | Days 1 and 8 of course 1 and then day 1 of course 2 (day 22)
  Comparison of pharmacokinetic parameters among the dose levels and drug-drug interaction performed using non-parametric statistical methods for K-independent samples.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wee Ma, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania